CLINICAL TRIAL: NCT06559709
Title: Implementing a Plant-Based Whole-Foods Meal Delivery Service for Patients Undergoing Autologous Hematopoietic Cell Transplantation for Multiple Myeloma: A Pilot Study
Brief Title: A Plant-Based Whole-Foods Meal Delivery Service for Patients With Multiple Myeloma Undergoing Autologous Hematopoietic Cell Transplant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: Swim Across America (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: RG1124594; NCI-2024-05448 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 20501 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2024-07-15; First posted 2024-08-19 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Specimen Handling; Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive care (meal delivery service) (Experimental): Patients receive 3 meals per day and snacks delivered twice weekly and meet with dietitian once weekly on days -7 to 28. Patients undergo blood and stool sample collection on study.
  Interventions: Procedure: Biospecimen Collection; Other: Dietary Intervention; Other: Medical Chart Review; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood and stool sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Other: Dietary Intervention — Receive 3 meals per day and snacks
  Other Names: Dietary Modification; intervention, dietary; Nutrition Intervention; Nutrition Interventions; Nutritional Interventions
Other: Dietary Intervention — Meet with dietitian
  Other Names: Dietary Modification; intervention, dietary; Nutrition Intervention; Nutrition Interventions; Nutritional Interventions
Other: Medical Chart Review — Ancillary studies
  Other Names: Chart Review
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial evaluates the impact of a plant-based whole-foods delivery service on the microbiome in patients with multiple myeloma undergoing an autologous hematopoietic cell transplant. An autologous hematopoietic cell transplant is a procedure in which blood-forming stem cells (cells from which all blood cells develop) are removed, stored, and later given back to the same person. Loss of microbial diversity within the intestinal tract has been associated with poor outcomes for patients receiving autologous stem cell transplantation. A plant-based whole meal delivery service may increase the intake of foods high in fiber and nutrients therefore improve microbial health during the peri-transplant period. In this pilot study, study investigators will explore the feasibility of this approach.

DETAILED DESCRIPTION:
OUTLINE:

Patients receive 3 meals per day and snacks delivered twice weekly and meet with dietitian once weekly on days -7 to 28. Patients undergo blood and stool sample collection on study.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent prior to initiation of any study procedures
* Planned first autologous stem cell transplantation for multiple myeloma
* Planned outpatient treatment for the duration of transplantation (if admitted, the investigators will request that caregivers bring the meals/snacks to the hospital as they might with other food prepared at home)
* Access to a refrigerator
* Ability to reheat foods
* Able to consume an oral diet at enrollment
* Able to communicate clearly regarding aspects of the study: e.g. Give feedback on logistics and meals, in order to maximize the operational data the investigators can gather in this pilot study
* At least 18 years of age

Exclusion Criteria:

* Major psychiatric diagnosis that impairs cognitive functioning or is not controlled at the time of the approach, as judged by the patient's medical team
* Planned inpatient transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2024-10-14 (Actual); Primary Completion 2025-08-29 (Actual); Study Completion 2025-08-29 (Actual)

PRIMARY OUTCOMES:
Enrollment rate | Up to 1 year
  The proportion of eligible patients who consent to enroll in the study will be computed based on the number approached and estimated with 95% confidence intervals. Reasons for non-participation will be summarized.
Collection rate | Up to 1 month post transplant
  Collection rate will be the percentage of stool samples, blood samples and surveys collected.
Tolerability of the delivered diet: Patient opinion | Up to 1 month post transplant
  Patient opinion of the delivered meals will be assessed using qualitative end-study surveys.
Tolerability of the delivered diet: Proportion of meals consumed | Up to 1 month post transplant
  Patient acceptability of the delivered meals will be assessed using proportions of the delivered meals consumed based on multi-day food diaries and 24-hour recall assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Kate Markey, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-08-07): https://cdn.clinicaltrials.gov/large-docs/09/NCT06559709/ICF_000.pdf